CLINICAL TRIAL: NCT01739920
Title: Comparative Efficacy of Two Different Regimens of Povidone-iodine 5% Eye Drops Instillation in Reducing Conjunctival Bacterial Flora
Brief Title: Comparative Efficacy of Different Regimens of PVPI 5% Eye Drops Instillation in Reducing Conjunctival Bacterial Flora
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Leticia Fernandes Barroso, MD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2516/2010; 2010/17350-6 (Other Grant/Funding Number: Fundação de Amparo à Pesquisa do Estado de São Paulo)
Record Dates: First submitted 2012-11-28; First posted 2012-12-04 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Eye Infections
Keywords: Povidone-Iodine; Ophthalmic Solutions; Endophthalmitis; Preoperative procedures
MeSH Terms: conditions — Eye Infections; Endophthalmitis | interventions — Povidone-Iodine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Povidone-iodine (Experimental): 1 drop of povidone-iodine 5% will be instilled at time zero, 20-minute and 28-minute study period.
  Interventions: Other: Povidone-iodine
- Povidone-iodine and Saline Solution (Active Comparator): 1 drop of saline solution 0.9% will be instilled at time zero and 20-minute. At 28-minute will be instilled 1 drop of Povidone-iodine 5%.
  Interventions: Other: Povidone-iodine; Other: Saline Solution

INTERVENTIONS:
Other: Povidone-iodine — Povidone iodine 5% drop will be instilled into conjunctival sac.
Other: Saline Solution — 1 drop of saline solution 0.9% will be instilled into conjunctival sac.
  Arms: Povidone-iodine and Saline Solution

SUMMARY:
The present study intends to assess the efficacy of 3 drops of 5% povidone-iodine (PVPI) eyedrops in reducing the bacterial flora in a conjunctival sac fundus compared to the standard procedure consisting of the application of 1 PVPI eyedrop 2 min before any intraocular surgical procedure.

DETAILED DESCRIPTION:
Studies have demonstrated that the external bacterial flora of the patients in most cases is the actual source of infection. The objective of antisepsis is to eliminate or significantly reduce the number of microorganisms in the surgical field at the time of surgery. The eyelids and the conjunctiva are considered to be quite common sources of bacteria that can lead to endophthalmitis. Thus, it is believed that by reducing the number and growth of bacteria on the ocular surface and adnexa before surgery, the risk of postoperative infection would be lower. Povidone-iodine 5% eye drops has been used in preoperative cataract surgery to prevent endophthalmitis and is the standard prophylactic action in preventing postoperative endophthalmitis being widely compared with other antibiotic eye drops and their associations. The standard procedure of prophylaxis of postoperative endophthalmitis corresponds to applying a single drop of povidone-iodine 2min before any intraocular surgical procedure. However, few studies have assessed the effectiveness of povidone-iodine 5% eye drops using different dosing regimens to achieve the best bactericidal effect. The aim of this study is to investigate different dosages with respect to the use of povidone-iodine drops to optimize the effectiveness of the agent, ensuring the best exogenous endophthalmitis prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* No systemic or ocular infection;
* Absence of auto-imune disease or immunosuppressive therapy;
* No use of systemic or topic antibiotics in the last 30 days;
* No previous ocular surgery or trauma in the study eye in the last 30 days;
* No history of allergy to povidone iodine;
* Signed informed consent.

Exclusion Criteria:

* Presence of blepharitis, ectropion, entropion, trichiasis or distichiasis;
* Diabetes Mellitus;
* Any systemic condition that, at the discretion of the investigators, would facilitate or contribute to infection, such as influenza;
* Inability to understand and sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Proportion of negative cultures after treatment in both groups | At 30-minute study period, a conjunctival sac swab will be obtained
  Conjunctival swab will be obtained five minutes before and 30 minutes after the first povidone iodine drop will be instilled into the conjunctival sac of study eye. Conjunctival swabs were incubated aerobically in enriched Thioglycolate liquid medium (meat broth) and in three solid culture media (Agar Chocolate, Trypticase Soy Agar with 5% sheep blood, and Agar Sabouraud).

SECONDARY OUTCOMES:
Difference in corneal thickness change between groups. | At 35-minute study period.
  Corneal paquimetry will be performed before and after procedure using OcuScan Alcon RXP (Alcon, Fortworth, Texas).

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Jorge, MD, PhD, Principal Investigator — University of Sao Paulo; Leticia F Barroso, MD, Principal Investigator — Clinics Hospital of Ribeirão Preto, School of Medicine of Ribeirão Preto, USP
Locations (1):
- Clinics Hospital of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil